CLINICAL TRIAL: NCT05667571
Title: A Mixed-Methods Pilot Study of Symptom Communication in Advanced Cancer: Patterns and Associating Factors
Brief Title: Symptom Communication in Advanced Cancer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201807052RINC
Record Dates: First submitted 2022-09-27; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2018-09

CONDITIONS: Communication; Cancer; Symptom, Behavioral
MeSH Terms: conditions — Communication; Neoplasms; Behavioral Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Improving patient-provider communication is a fundamental and cost-effective method to advance patient outcomes, including symptom management which is often the primary goal of care for patients with advanced cancer. Unfortunately, some studies revealed the poor quality of symptom communication among cancer patients and healthcare providers. While these evidences suggest important gaps in communication about symptoms with some of the most vulnerable patients, little is known about the patterns and associating factors of symptom communication.

Purpose and Specific Aims The proposed 3-year pilot project aims to provide an enrich and systematic description of symptom communication by validating a newly developed typology of interaction patterns of symptom communication (TIPSC) between patients with advanced cancer, their caregivers, and healthcare providers and explore factors related to each interaction pattern. The specific aims are to: (1) validate TIPSC in Taiwanese advanced cancer population, (2) explore patients' /caregivers' experience and thoughts of symptom discussion in regard to their interaction patterns and symptom management, and (3) examine relationships between interaction patterns and (a) demographic factors, (b) symptom severity, (c) congruence in symptom assessment between patients/caregivers and providers, (d) patients'/caregivers' perceived ability to communicate with providers, and (e) patient/caregiver satisfaction.

Sampling This pilot study plans to recruit about 50 patient/caregiver - oncologist dyads. The recruitment process contains three stages. First, medical oncologists who are currently in clinical practice at participating institutions and care for patients with solid tumors will be approached. Second, participating oncologists' patients will be recruited if they are: (1) currently a patient of a participating oncologist, (2) diagnosed with stage III or IV solid cancer, (3) aged 20 years or older, (4) able to tolerate an interview that will last approximately 30 minus, and (5) able to speak Chinese or Taiwanese. Finally, if applicable, adult caregivers who intent to join selected out-patient-department (OPD) visit with the patients will also be recruited.

Research Design This is a mixed-methods study with a two-phase exploratory sequential design. The first phase is a qualitative descriptive study in which the investigators will record patient/caregiver-oncologist OPD visits and conduct patient/caregiver interviews to address aim 1 and 2. Discourse and conversation analysis will be used to analyze the recorded visits and content analysis will be used to analyze the interviews. The second phase is a correlational study in which the investigators use questionnaires to measure variables and examine their relationship with interaction patterns (aim 3). Descriptive statistics, binomial logistic regression, and linear regression will be used to analyze quantitative data.

Expecting Results This is a pioneering study addressing the patterns and associating factors of symptom communication in Taiwanese patients with advanced cancer. The findings will systematically map out the patient/caregiver-provider symptom communication and identify relationships between communication patterns and meaningful indicators. This proposed study is a critical step to understand patient/caregiver-provider communication regarding symptoms in order to pinpoint symptom management and communication barriers and design proper interventions in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Currently a patient of a participating physician
* Diagnosed with advanced solid cancer (TNM stage III or IV)
* Aged 20 years or older
* Able to tolerate an interview that will last approximately 30 minus
* Able to speak Chinese or Taiwanese.

Exclusion Criteria:

* Do not experience any symptoms
* Are hospitalized at recruitment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Chinese Patients' Satisfaction Scale (C-PSS) | Once, immediately after outpatient visit
  patient satisfaction

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer (EORCT-QLQ C30) | Once, immediately after outpatient visit
  congruence of symptom management between patients and providers

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05667571/Prot_SAP_000.pdf